CLINICAL TRIAL: NCT02935504
Title: PRogram In Support of Moms (PRISM): A Pilot Group Randomized Controlled Trial
Brief Title: PRogram In Support of Moms (PRISM): A Pilot Study
Acronym: PRISM-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nancy Byatt, Associate Professor of Psychiatry and Obstetrics & Gynecology, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H00004195; UL1TR000161 (NIH)
Record Dates: First submitted 2016-10-04; First posted 2016-10-17 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Perinatal Depression
Keywords: Depression; Pregnancy; Postpartum
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Program In Support of Moms PRISM (Experimental): PRISM includes MCPAP for Moms and training, implementation support, and toolkits for Ob/Gyn practices on depression screening, assessment and treatment.
  Interventions: Behavioral: PRogram In Support of Moms (PRISM)
- MCPAP for Moms (Active Comparator): Consists of access to psychiatric consultation and resources and referrals through MCPAP for Moms - MCPAP for Moms is available free of charge to all Ob/Gyn practices in Massachusetts.
  Interventions: Behavioral: MCPAP for Moms

INTERVENTIONS:
Behavioral: PRogram In Support of Moms (PRISM) — PRISM Intervention Provider and staff training Webinar Delivered in person Engage providers - Registered Nurses (RN) and Patient Care Assistants (PCA) and ensure they attend:
  Toolkit Care coordination Psychiatric consultation Implementation support
  1. Engage clinic leaders and staff
  2. Identify leadership group and prepare for change
  3. Assess readiness to implement PRISM
  4. Identify steps to achieve goals
  5. Implement PRISM components into the clinic
  6. Support, encourage and sustain change Office prompts Screening procedures Plus all MCPAP for Moms intervention
  Other Names: Rapid Access to Perinatal Psychiatric care in Depression; RAPPID
  Arms: Program In Support of Moms PRISM
Behavioral: MCPAP for Moms — MCPAP for Moms Provider and staff training Delivered via web RN and PCA admin staff recommended to attend 30-60 minute presentation on perinatal depression Access to telephonic psychiatric consultation with MCPAP for Moms perinatal psychiatrist for Ob/Gyns Access to one-time face-face evaluation with patient by a MCPAP for Moms psychiatrist for assessment and treatment recommendations for Ob/Gyn provider Access to Provider Toolkit which includes assessment and treatment protocols (available at www.mcpapformoms.org) Resource provision/referrals
  Arms: MCPAP for Moms

SUMMARY:
The primary goal of this study is to evaluate the PRogram In Support of Moms (PRISM) that aims to improve women's access to and participation in perinatal depression treatment and thereby improve depression outcomes

DETAILED DESCRIPTION:
Major depressive disorder continues to be the leading cause of disability among women of reproductive age and major public health concern. Upwards of 1 in 5 women suffer from depression during pregnancy or within a year after giving birth. It has negative effects on birth outcomes, infant attachment, behavior and development. Maternal suicide causes 20% of postpartum deaths in depressed women. Although the majority of women are amenable to depression screening, screening alone does not improve treatment entry or outcome. Despite the availability of effective evidence-based treatments and frequent contact with obstetric providers, less than one-third of women who screen positive for depression receive treatment. Ob/Gyn practices need supports in place to adequately address depression in their patient populations. Thus, the Investigators developed a program called "PRogram In Support of Moms" (PRISM) that aims to leverage existing roles and resources to target patient, provider, and system level barriers to perinatal depression treatment. PRISM aims to improve perinatal depression treatment and treatment response rates through: (1) access to psychiatric telephone consultation for Ob/Gyn providers; (2) clinic-specific implementation of stepped care, including training support and toolkits; and, (3) proactive treatment engagement, patient monitoring, and stepped treatment response to depression screening/assessment. Four practices were randomly assigned to PRISM versus an active comparison group called MCPAP for Moms which is a state-wide telephonic perinatal psychiatry program. The Investigators will compare the effectiveness of PRISM vs. MCPAP for Moms to improve depression severity and treatment participation in pregnancy through 3 months postpartum among patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 18-55 years
3. English speaking
4. 4-36 weeks gestational age (GA) or 2-12 weeks postpartum
5. Receiving care from one of the 4 participating clinics (2 clinics which will participate in PRISM and 2 with access to MCPAP for Moms)
6. Edinburgh Postnatal Depression Scale score (EPDS) ≥10
7. Able to communicate in written and spoken English; and
8. Cognitively able to participate in informed consent

Exclusion Criteria:

1. Lack of verbal and written English fluency
2. Under age 18 or over age 55
3. Current active substance use disorder
4. Bipolar disorder diagnosis as determined by the Mini-international Neuropsychiatric Interview (M.I.N.I.)
5. Psychotic component to illness as determined by the M.I.N.I.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Depression Severity | Baseline to 10-35 weeks follow-up
  To compare changes in depression severity as measured by Edinburgh Postnatal Depression Scale (EPDS) from baseline to follow-up (10-35 weeks) among pregnant and postpartum women in PRISM versus MCPAP for Moms.

SECONDARY OUTCOMES:
Provider Fidelity | Baseline to 1 year follow-up (post intervention)
  To determine change in knowledge, attitudes, and practices as measured by S-KAP toward depression screening and treatment from baseline (pre implementation) to 1 year follow-up (post implementation) among providers in PRISM versus MCPAP for Moms practices.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Byatt, DO, MS, MBA, Principal Investigator — • UMass Memorial Medical Center/UMass Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Switzerland: Department of Health Statistics and Informatics; Information EaRCotWHO. The Global Burden of Disease: 2004 update; 2008.
- [Background] Grote NK, Bridge JA, Gavin AR, Melville JL, Iyengar S, Katon WJ. A meta-analysis of depression during pregnancy and the risk of preterm birth, low birth weight, and intrauterine growth restriction. Arch Gen Psychiatry. 2010 Oct;67(10):1012-24. doi: 10.1001/archgenpsychiatry.2010.111. PMID 20921117
- [Background] Paulson JF, Keefe HA, Leiferman JA. Early parental depression and child language development. J Child Psychol Psychiatry. 2009 Mar;50(3):254-62. doi: 10.1111/j.1469-7610.2008.01973.x. Epub 2008 Oct 23. PMID 19175819
- [Background] Deave T, Heron J, Evans J, Emond A. The impact of maternal depression in pregnancy on early child development. BJOG. 2008 Jul;115(8):1043-51. doi: 10.1111/j.1471-0528.2008.01752.x. PMID 18651886
- [Background] Lindahl V, Pearson JL, Colpe L. Prevalence of suicidality during pregnancy and the postpartum. Arch Womens Ment Health. 2005 Jun;8(2):77-87. doi: 10.1007/s00737-005-0080-1. Epub 2005 May 11. PMID 15883651
- [Background] Carter FA, Carter JD, Luty SE, Wilson DA, Frampton CM, Joyce PR. Screening and treatment for depression during pregnancy: a cautionary note. Aust N Z J Psychiatry. 2005 Apr;39(4):255-61. doi: 10.1080/j.1440-1614.2005.01562.x. PMID 15777362
- [Background] Kozhimannil KB, Adams AS, Soumerai SB, Busch AB, Huskamp HA. New Jersey's efforts to improve postpartum depression care did not change treatment patterns for women on medicaid. Health Aff (Millwood). 2011 Feb;30(2):293-301. doi: 10.1377/hlthaff.2009.1075. PMID 21289351
- [Background] Gilbody S, Sheldon T, House A. Screening and case-finding instruments for depression: a meta-analysis. CMAJ. 2008 Apr 8;178(8):997-1003. doi: 10.1503/cmaj.070281. PMID 18390942
- [Background] Yonkers KA, Smith MV, Lin H, Howell HB, Shao L, Rosenheck RA. Depression screening of perinatal women: an evaluation of the healthy start depression initiative. Psychiatr Serv. 2009 Mar;60(3):322-8. doi: 10.1176/appi.ps.60.3.322. PMID 19252044
- [Background] Weissman MM, Pilowsky DJ, Wickramaratne PJ, Talati A, Wisniewski SR, Fava M, Hughes CW, Garber J, Malloy E, King CA, Cerda G, Sood AB, Alpert JE, Trivedi MH, Rush AJ; STAR*D-Child Team. Remissions in maternal depression and child psychopathology: a STAR*D-child report. JAMA. 2006 Mar 22;295(12):1389-98. doi: 10.1001/jama.295.12.1389. PMID 16551710
- [Background] Smith MV, Shao L, Howell H, Wang H, Poschman K, Yonkers KA. Success of mental health referral among pregnant and postpartum women with psychiatric distress. Gen Hosp Psychiatry. 2009 Mar-Apr;31(2):155-62. doi: 10.1016/j.genhosppsych.2008.10.002. Epub 2008 Dec 3. PMID 19269536
- [Background] Marcus SM, Flynn HA, Blow FC, Barry KL. Depressive symptoms among pregnant women screened in obstetrics settings. J Womens Health (Larchmt). 2003 May;12(4):373-80. doi: 10.1089/154099903765448880. PMID 12804344
- [Background] Rowan P, Greisinger A, Brehm B, Smith F, McReynolds E. Outcomes from implementing systematic antepartum depression screening in obstetrics. Arch Womens Ment Health. 2012 Apr;15(2):115-20. doi: 10.1007/s00737-012-0262-6. Epub 2012 Mar 1. PMID 22382279
- [Background] Byatt N, Levin LL, Ziedonis D, Moore Simas TA, Allison J. Enhancing Participation in Depression Care in Outpatient Perinatal Care Settings: A Systematic Review. Obstet Gynecol. 2015 Nov;126(5):1048-1058. doi: 10.1097/AOG.0000000000001067. PMID 26444130
- [Derived] McNicholas E, Boama-Nyarko E, Julce C, Nunes AP, Flahive J, Byatt N, Moore Simas TA. Understanding Perinatal Depression Care Gaps by Examining Care Access and Barriers in Perinatal Individuals With and Without Psychiatric History. J Womens Health (Larchmt). 2023 Oct;32(10):1111-1119. doi: 10.1089/jwh.2022.0306. Epub 2023 Aug 16. PMID 37582274